CLINICAL TRIAL: NCT04176666
Title: NettOpp: The Development and Evaluation of an App-based Selective Intervention for Adolescents Exposed to Cyberbullying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Principal Investigator, Henriette Kyrrestad, Associate Professor, University of Tromso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 161212 NettOpp - effektstudie; 545417 (Other: NSD - Norwegian Centre for Research Data)
Record Dates: First submitted 2019-11-14; First posted 2019-11-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cyberbullying
Keywords: cyberbullying; cyberaggression; mobile application
MeSH Terms: conditions — Cyberbullying

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group receiving NettOpp (Experimental): The effectiveness study will be conducted as a randomized controlled trial with an intervention group and a waiting-list control group. Data will be collected at baseline (T1, pre intervention) and after about 2 weeks of intervention (T2, post intervention). A follow-up evaluation (T3) will be conducted after about 3 months to examine if the effects were stable over time.
  Interventions: Device: NettOpp
- Control group (No Intervention): The control group will receive the intervention after study completion.

INTERVENTIONS:
Device: NettOpp — NettOpp is a mobile application for adolescents aged 11-16 years who have been exposed to cyberbullying or cyberaggression.
  Arms: Intervention group receiving NettOpp

SUMMARY:
The aim of the project is to develop and evaluate an app-based intervention for adolescents who have been exposed to cyberbullying. The overarching goal is to offer a low-threshold intervention, called NettOpp, that is easy accessible and free to use for every junior high school student who has experienced cyberbullying in Norway.

DETAILED DESCRIPTION:
The main aim of the intervention is to increase coping strategies for adolescents who have been exposed to cyberbullying. More specifically the aims are to increase 1) knowledge about cyberbullying, 2) help-seeking behavior, 3) coping strategies with cyberbullying, 4) to reduce mental health problems, and 5) cyberbullying, and 6) to increase self-esteem and the 7) sleeping quality of the adolescents.

To evaluate the mobile application three studies will be conducted: A lab test, a pilot study, and a larger effectiveness study with a follow-up examination after 3 months. The lab test will be conducted to examine the quality of the prototype of the app in order to find out if adjustments have to be made. Thereafter, a pilot study will be conducted with adolescents that were exposed to cyberbullying in the past six months. The pilot study will use a pre-post design.The effectiveness study will be conducted as a randomized controlled trial with an intervention group and a waiting-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents whose guardians have given consent and who agree to take part in the study

Exclusion Criteria:

* severe developmental or cognitive challenges

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 709 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
SDQ (Strengths and Difficulties Questionnaire) | From baseline to 2 weeks after intervention, and after 3 months as follow-up.
  Adolescents: SDQ (Goodman, 1997): A 25 item self-report assessing mental health and psychosocial functioning in 11-17 years old adolescents on a three point scale.
CATS (Child and Adolescent Trauma Screening) | From baseline to 2 weeks after intervention, and after 3 months as follow-up.
  Adolescents: CATS (Sachser et al., 2017): A 20 item self-report assessing posttraumatic stress-symptoms for 7-17 year old adolescents on a four point scale.
WHO-5 (WHO-Five Well-being Index) | From baseline to 2 weeks after intervention, and after 3 months as follow-up.
  Adolescents: WHO-5 (WHO, 1998): A five item self-report questionnaire assessing well-being on a six point scale.

SECONDARY OUTCOMES:
Help-seeking behavior | From baseline to 2 weeks after intervention, and after 3 months as follow-up.
  Adolescents: three self-report items measuring if they sought help, who they sought help from, and if they received the help they needed.
Cyberbullying | From baseline to 2 weeks after intervention, and after 3 months as follow-up.
  Adolescents: Cyberbullying (Olweus, 1993): One self-report item measuring the frequency of cyberbullying exposure.
Self-liking and Competence Scale | From baseline to 2 weeks after intervention, and after 3 months as follow-up.
  Adolescents: Self-liking and Competence Scale (Silvera, Neilands, & Perry, 2001; Tafarodi & Swann, 2001): A 20 item self-report assessing self-liking and self-competence.
Sleeping quality | From baseline to 2 weeks after intervention, and after 3 months as follow-up.
  Adolescents: Sleeping quality will be measured with six questions with different response categories from the Bergen Child Study (Hysing, Harvey, Stormark, Pallesen, & Sivertsen, 2018).
CCQ (Cyberbullying Coping Questionnaire) | From baseline to 2 weeks after intervention, and after 3 months as follow-up.
  Adolescents: CCQ (Jacobs, Völlink, Dehue, & Lechner, 2015): A 17 item self-report assessing how often the adolescents use the different cyberbullying coping strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Henriette Kyrrestad, PhD, Principal Investigator — UiT The Arctic University of Norway
Locations (1):
- UiT The Arctic University of Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaiser S, Martinussen M, Adolfsen F, Breivik K, Kyrrestad H. An App-Based Intervention for Adolescents Exposed to Cyberbullying in Norway: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Nov 8;10(11):e31789. doi: 10.2196/31789. PMID 34747704